CLINICAL TRIAL: NCT05996276
Title: Impact of Dose to Cardiac Substructures on Survival in Patients With Esophageal Cancer Treated With Radiotherapy or Chemoradiotherapy
Brief Title: Impact of Dose to Cardiac Substructures on Survival in Patients With Esophageal Cancer Treated With Radiotherapy or Chemoradiotherapy (SATIATION)
Acronym: SATIATION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0144 - SATIATION
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2023-08

CONDITIONS: Esophagus Cancer
Keywords: radiotherapy; cardiotoxicity
MeSH Terms: conditions — Esophageal Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Treatment of non-operable esophageal cancers is based on radiochemotherapy, or exclusive radiotherapy.

The cardiac toxicity of radiotherapy in the treatment of thoracic tumor localizations is well documented, however, more and more studies are calling for the use of dosimetric parameters related to cardiac sub-structures to be integrated into clinical practice, rather than considering the heart as a whole.

With this in mind, the aim of this study is to define the parameters, particularly dosimetric ones linked to cardiac sub-structures, influencing survival in patients treated with exclusive radiotherapy or radiochemotherapy for esophageal cancer.

DETAILED DESCRIPTION:
Treatment of non-operable esophageal cancers is based on radiochemotherapy, or exclusive radiotherapy.

The cardiac toxicity of radiotherapy in the treatment of thoracic tumor localizations is well documented, however, more and more studies are calling for the use of dosimetric parameters related to cardiac sub-structures to be integrated into clinical practice, rather than considering the heart as a whole.

Although most of these data have been studied in populations with long-term follow-up, such as breast cancer, cardiac toxicity and the reduced survival it entails are also found in diseases such as esophageal cancer.

With this in mind, the aim of this study is to define the parameters, particularly dosimetric ones linked to cardiac sub-structures, influencing survival in patients treated with exclusive radiotherapy or radiochemotherapy for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically or cytologically proven esophageal cancer
* Localized or locally advanced esophageal cancer treated with radiochemotherapy or exclusive radiotherapy
* Tumor dose ≥ 50 Gy
* Non-opposition of living patients formulated
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Age < 18 years
* Patient treated with upfront surgery
* Tumor dose < 50 Gy
* Other concomitant neoplasia
* Metastatic patient
* Refusal to participate
* Patient under legal protection (guardianship, curatorship, etc...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-operated adult patients with localized or locally advanced esophageal cancer treated with radiochemotherapy or radiotherapy alone for curative purposes.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | through study completion, an average of 1 year
  OS is defined as the time elapsed between inclusion and death, whatever the cause.

SECONDARY OUTCOMES:
The rate of cardiac events. | through study completion, an average of 1 year
  The rate of cardiac events.
Response rate. | through study completion, an average of 1 year
  Response rate.
Progression-free survival (PFS). | through study completion, an average of 1 year
  PFS is defined as the time elapsed between inclusion and tumor progression assessed by an expert panel according to RECIST v1.1 criteria, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Bourbonne, MD, PhD, Principal Investigator — Radiation Oncology Department, Brest University Hospital
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement